CLINICAL TRIAL: NCT06688344
Title: Effectiveness of Focused Extracorporeal Shock Wave Therapy Applied as an Addition to Conventional Physiotherapy Program After Anterior Cruciate Ligament Reconstruction
Brief Title: Efficacy of Focused Extracorporeal Shock Wave Therapy After Anterior Cruciate Ligament Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Berivan Beril Kılıç (Other)
Responsible Party: Sponsor-Investigator, Berivan Beril Kılıç, assistant professor, Biruni University
Organization: Biruni University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2982164
Record Dates: First submitted 2024-11-11; First posted 2024-11-14 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: ACL Reconstruction; Extracorpereal Shock Wave Therapy
Keywords: Physiotherapy and rehabilitation; ESWT; ACL reconstruction
MeSH Terms: interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): fESWT
  Interventions: Other: fESWT; Other: Conventional Physiotherapy
- Control group (Sham Comparator)
  Interventions: Other: Conventional Physiotherapy; Other: shamfESWT

INTERVENTIONS:
Other: fESWT — fESWT will be applied for 1 session between weeks 4-9. The device will be set to low intensity at 0.20 mJ/mm2 - 4 Hz, 500 pulses will be applied from the tibiofemoral interval to the center of the tibiofemoral joint, and 1000 pulses will be applied to the soft tissues around the patella.
  Arms: Intervention group
Other: Conventional Physiotherapy — Participants will be included in the traditional physiotherapy program for the first 9 weeks, and exercise progression will be provided in the form of weekly checks in the 10-12 week period. Between the 12-24th weeks, the exercise program will continue with face-to-face follow-up twice a month.
  The traditional physiotherapy program to be applied in the first 9-week period will be as follows :
  Week 1 Weight Transfer as Tolerable, NMES, Elevation, Cold Application, Ankle Pumping Exercises, Heel Slide Exercises, Isometric Quadriceps Exercises, Straight Leg Raise Exercises, Extension Brace
  Week 2-3 Weight Transfer, Gait Training, NMES, Heel Slide Exercises, Straight Leg Raise, Quadriceps and Adductor Isometric Exercises, Extension Brace, Bicycle, Hip Abduction-Adduction Exercises
  Week 4-8. week Mini Squat, Leg Press, Soft Ground Walking, Neuromuscular Training on Balance Board, Functional Strengthening with Elastic Band, Stair Climbing Up and Down
  Other Names: Rehabilitation
Other: shamfESWT — Participants in the control group will receive sham fESWT once a week in weeks 4-9. Participants will be prepared in the same way as the fESWT procedure, but the application will be done with a sham device.
  Arms: Control group

SUMMARY:
The aim of this clinical trial is to determine the effectiveness of fESWT in rehabilitation after ACL reconstruction. The main questions it aims to answer are:

Is fESWT applied in addition to conventional physiotherapy effective in physiotherapy-related parameters?

Researchers will compare conventional physiotherapy and conventional physiotherapy + fESWT to see if fESWT provides benefits in addition to conventional physiotherapy.

Participants:

They will receive the conventional physiotherapy program 2 days per week. In addition, the intervention group will receive low-intensity fESWT 1 day per week.

Participants' muscle strength, postural balance, range of motion, pain scores and functional status will be assessed.

DETAILED DESCRIPTION:
Extracorporeal shock wave therapy (ESWT) is a safe, effective and non-invasive treatment option that can be used in different pathologies of the musculoskeletal system. It is based on the production of acoustic waves that interact directly with cells through mechanotransduction and activate the metabolic process that leads to tissue remodeling. ESWT can be classified as focused ESWT (fESWT) and radial ESWT (rESWT). While rESWT has a more superficial effect and reaches the maximum energy at the skin surface and distributes it radially to the tissue, fESWT develops the maximum energy at a focus located deeper in the body tissues. Studies have suggested that ESWT can be applied in combination with physiotherapy in patients affected by musculoskeletal disorders . In the literature, its effectiveness has been investigated in different musculoskeletal problems such as lateral epicondylitis, rotator cuff tendinopathy, Achilles tendinopathy, patellar tendinopathy, greater trochanteric pain syndrome, plantar fasciitis, and the best evidence supporting the use of ESWT has been obtained with low to medium energy levels for tendon disorders and high energy levels for tendon calcification and bone pathologies . The usability of ESWT treatment in knee-related pathologies has been discussed in the literature. In the treatment of ligament injuries such as the medial collateral ligament, fESWT has been shown to be a reliable and safe light energy shock wave treatment for the management of injuries without surgical indications . It has been reported that it is useful for inducing neovascularization in knee tendon injuries, improving blood flow in the bone-tendon junction, and supporting tissue repair. It has been thought that it has chondroprotective, anti-inflammatory, neovascularization, antiapoptotic and tissue regeneration effects on tissues, and therefore can be used in osteoarthritis. Another situation where the effect of ESWT on knee pathologies has been investigated is anterior cruciate ligament (ACL) surgeries. ACL reconstruction surgery aims to restore knee functions by providing the tightest possible repair so that the reconstruction of the torn ligament can be an excellent biological replacement. The functional outcome of this surgery depends on the solid healing of the graft-bone union in the bone tunnel. It is known that if the bone and tendon do not heal together, this may lead to knee pathology in the future. Although the studies on the use of ESWT after ACL surgery are quite limited, more focus has been placed on the effect of ESWT on the graft. Wang et al. applied 1 session of fESWT in operating room conditions during anterior cruciate ligament reconstruction surgery and reported that the patients had higher functional levels compared to the control group at 1 and 2 years. Song et al. included 72 patients who underwent anterior cruciate ligament reconstruction and applied ESWT once a week starting from the 2nd postoperative day in addition to the standard physiotherapy protocol for 6 weeks. Significant improvements in 6-week functionality and range of motion values compared to the control group, and no significant difference was found between the groups at the end of 6 months. Moi et al. compared graft healing and knee functional results in groups that received only physiotherapy, physiotherapy + ESWT once a week between weeks 6-8, and ESWT once a week between weeks 7-12. As a result, they reported that 6-session application had positive effects on graft healing; and there was no difference between knee functional scores at the end of 6 months . In another study, Weninger et al. applied ESWT at 1 and 6 weeks and evaluated the patients at 3, 6, 9 and 12 months. They reported that there were greater improvements in knee functionality, daily living and pain scores at all times in the ESWT group compared to the control group in the evaluation parameters. In addition, they reported that graft maturation was better in the ESWT group . Rehabilitation protocols commonly used after surgery aim to restore mobility and regain independence in daily living activities through muscle strengthening, functional exercises and proprioception training. When the studies conducted after anterior cruciate ligament surgery in the literature are examined, the effects of ESWT on outcomes such as muscle strength, proprioception and postural stability, which are targeted to be increased with rehabilitation protocols, have not been examined. No studies have been found in the literature examining the effects of ESWT on muscle strength, range of motion and postural stability, which are affected after surgery and targeted to be improved in the rehabilitation program, other than the effect of ESWT on graft healing after ACL reconstruction surgery. In this context, the aim of this study is to investigate the effects of fESWT applied in addition to the traditional rehabilitation protocol after anterior cruciate ligament surgery on muscle strength, range of motion, postural stability, pain and functionality.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45 years
* Unilateral ACL rupture
* Isolated ACL injury
* Hamstring graft

Exclusion Criteria:

* Previous knee injury and anterior cruciate ligament revision
* Synovitis, stiffness, tension
* History of systemic diseases such as rheumatoid arthritis, osteoarthritis, osteoporosis
* Presence of tumor
* Deep vein thrombosis or vascular pathology in the lower extremity
* RA or accompanying comorbidities
* Having had intra-articular injection within 6 months
* Cognitive impairment

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Knee extansor muscle strength | a time frame of 6,9,12 weeks
  The strength of the participants' knee flexor and knee extensor muscles will be measured with a hand held dynamometer.
  Knee extensor muscle strength will be performed in a sitting position. Participants will be seated on an examination table with their knees bent at 60° and their feet off the ground. The dynamometer will be placed on the front of the distal tibia, just above the malleoli for extensor strength and the posterior aspect of the distal tibia, just above the malleoli for flexor strength . Participants will grip the examination table with their hands for stabilization and will be asked to apply force to the dynamometer for 5 seconds with maximum force. 3 repetitions will be performed and the average will be calculated by dividing by body weight in N/kg.
postural stability | a time frame of 6,9,12 weeks
  Participants' single-leg and double-leg postural stability assessments will be performed with the Biodex brand balance system. General balance index (OSI), anteroposterior balance index (APSI) and mediolateral balance index (MLSI) will be recorded. Measurements will be performed without shoes, with eyes open and arms crossed over the body. While the level of the system drops from 12 to 10 in the double-leg assessment, it will drop from 12 to 10 in the single-leg assessment. Participants will proceed to the test protocol consisting of 3 2o seconds each after a single trial measurement. The average score from the three test assessments will be calculated and recorded. 5-minute rest breaks will be given between the tests.

SECONDARY OUTCOMES:
range of motion | a time frame of 6,9,12 weeks
  Knee extension and flexion joint range of motion will be performed in the prone position with the help of a goniometer. Measurements will be repeated 3 times and the average will be recorded.
pain assessment - VAS | a time frame of 6,9,12 weeks
  The degree of pain of the participants will be assessed with a visual analog scale. Participants will be asked to give a value between 0-100 for the pain they feel in their knees and this score will be recorded. '0' means no pain is felt, while 100 means maximum pain is felt.
pain assessment-algometer | a time frame of 6,9,12 weeks
  Another method to be used in pain assessment is to evaluate the pain pressure threshold of the participants with an algometer. In the assessment to be made with an algometer, the previous research was taken as a reference for the reference measurement points. Accordingly, the reference points are - 10 cm lateral to the middle point of the upper edge of the patella, - 3 cm medial to the upper middle point of the patella, - the middle point between the lower edge of the patella and the tibial tuberosity, - 3 cm proximal to the upper edge of the patella - 3 cm medial to the tuberosity of the tibia at the pes anserinus insertion. Three 10-second assessments will be performed with a 30-second rest at each point and the average (Kg) value will be recorded for analysis.
Functionality and daily living activity assessment-IKDC | a time frame of 6,9,12 weeks
  IKDC (International Knee Documentation Committee): The IKDC Subjective Knee Form is designed to measure symptoms of various knee disorders such as ligament, meniscus and cartilage injuries and patellofemoral pain, and limitations in function and sports activities. It consists of 18 questions and 3 subscales. There are 7 questions for symptoms, 10 questions for sports activities and 1 question for function assessment. The total score range on the form varies between 0-100, with higher scores indicating fewer symptoms and a higher functional level. Its cultural adaptation was made by Çelik et al.
Functionality and daily living activity assessment-Lysholm Scale | a time frame of 6,9,12 weeks
  The scale, consisting of 8 questions, was designed to evaluate the results of knee ligament surgery, especially instability symptoms, in patients with anteromedial, anterolateral, combined anteromedial/anterolateral, posterolateral rotator knee ligament injuries or straight posterior instability. Scoring is done out of 100. Scores between 95-100 are considered excellent, 84-94 good results, 65-83 moderate and values below 65 poor results. The scale has been validated in Turkish.
Kinesiophobia assessment | a time frame of 6,9,12 weeks
  A scale consisting of 17 questions developed to assess the fear of pain associated with movement in patients with musculoskeletal pain. It includes occupational injury, re-injury and fearful avoidance parameters. The validity and reliability of the questionnaire in Turkish has been performed. The scale can be scored between 17 and 68. As the score on the scale increases, the level of kinesiophobia increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Faculy of Medicine-Department of Sports Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Tampa Kinezyofobi Ölçeği'nin Türkçe versiyonu ve test-tekrar test güvenirliği.
- [Result] Hapidou EG, O'Brien MA, Pierrynowski MR, de Las Heras E, Patel M, Patla T. Fear and Avoidance of Movement in People with Chronic Pain: Psychometric Properties of the 11-Item Tampa Scale for Kinesiophobia (TSK-11). Physiother Can. 2012 Summer;64(3):235-41. doi: 10.3138/ptc.2011-10. PMID 23729957
- [Result] Celik D, Coskunsu D, Kilicoglu O. Translation and cultural adaptation of the Turkish Lysholm knee scale: ease of use, validity, and reliability. Clin Orthop Relat Res. 2013 Aug;471(8):2602-10. doi: 10.1007/s11999-013-3046-z. Epub 2013 May 11. PMID 23666590
- [Result] Lysholm J, Gillquist J. Evaluation of knee ligament surgery results with special emphasis on use of a scoring scale. Am J Sports Med. 1982 May-Jun;10(3):150-4. doi: 10.1177/036354658201000306. PMID 6896798
- [Result] Celik D, Coskunsu D, KiliCoglu O, Ergonul O, Irrgang JJ. Translation and cross-cultural adaptation of the international knee documentation committee subjective knee form into Turkish. J Orthop Sports Phys Ther. 2014 Nov;44(11):899-909. doi: 10.2519/jospt.2014.4865. Epub 2014 Oct 16. PMID 25323139
- [Result] Medial patellofemoral ligament rekonstrüksiyonu sonrası kalça abduktör kas kuvvetlendirme egzersizlerinin diz fonksiyonu üzerine etkisi.
- [Result] Irrgang JJ, Anderson AF, Boland AL, Harner CD, Kurosaka M, Neyret P, Richmond JC, Shelborne KD. Development and validation of the international knee documentation committee subjective knee form. Am J Sports Med. 2001 Sep-Oct;29(5):600-13. doi: 10.1177/03635465010290051301. PMID 11573919
- [Result] Akbari A, Ghiasi F, Mir M, Hosseinifar M. The Effects of Balance Training on Static and Dynamic Postural Stability Indices After Acute ACL Reconstruction. Glob J Health Sci. 2015 Jul 31;8(4):68-81. doi: 10.5539/gjhs.v8n4p68. PMID 26573034
- [Result] Martin-Alguacil JL, Arroyo-Morales M, Martin-Gomez JL, Lozano-Lozano M, Galiano-Castillo N, Cantarero-Villanueva I. Comparison of knee sonography and pressure pain threshold after anterior cruciate ligament reconstruction with quadriceps tendon versus hamstring tendon autografts in soccer players. Acta Orthop Traumatol Turc. 2019 Jul;53(4):260-265. doi: 10.1016/j.aott.2019.04.012. Epub 2019 Jun 12. PMID 31201076
- [Result] Luc-Harkey BA, Safran-Norton CE, Mandl LA, Katz JN, Losina E. Associations among knee muscle strength, structural damage, and pain and mobility in individuals with osteoarthritis and symptomatic meniscal tear. BMC Musculoskelet Disord. 2018 Jul 27;19(1):258. doi: 10.1186/s12891-018-2182-8. PMID 30049269
- [Result] Sık Yapılan Ortopedik Ameliyatlar ve Rehabilitasyon Yaklaşımları. İstanbul Tıp Kitabevleri
- [Result] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Result] Rahim M, Ooi FK, Shihabudin MT, Chen CK, Musa AT. The Effects of Three and Six Sessions of Low Energy Extracorporeal Shockwave Therapy on Graft Incorporation and Knee Functions Post Anterior Cruciate Ligament Reconstruction. Malays Orthop J. 2022 Mar;16(1):28-39. doi: 10.5704/MOJ.2203.005. PMID 35519531
- [Result] Song Y, Che X, Wang Z, Li M, Zhang R, Wang D, Shi Q. A randomized trial of treatment for anterior cruciate ligament reconstruction by radial extracorporeal shock wave therapy. BMC Musculoskelet Disord. 2024 Jan 13;25(1):57. doi: 10.1186/s12891-024-07177-8. PMID 38216944
- [Result] Wang CJ, Ko JY, Chou WY, Hsu SL, Ko SF, Huang CC, Chang HW. Shockwave therapy improves anterior cruciate ligament reconstruction. J Surg Res. 2014 May 1;188(1):110-8. doi: 10.1016/j.jss.2014.01.050. Epub 2014 Jan 31. PMID 24560350
- [Result] Weninger P, Thallinger C, Chytilek M, Hanel Y, Steffel C, Karimi R, Feichtinger X. Extracorporeal Shockwave Therapy Improves Outcome after Primary Anterior Cruciate Ligament Reconstruction with Hamstring Tendons. J Clin Med. 2023 May 9;12(10):3350. doi: 10.3390/jcm12103350. PMID 37240456
- [Result] Wang CJ, Wang FS, Yang KD, Weng LH, Sun YC, Yang YJ. The effect of shock wave treatment at the tendon-bone interface-an histomorphological and biomechanical study in rabbits. J Orthop Res. 2005 Mar;23(2):274-80. doi: 10.1016/j.orthres.2004.07.004. PMID 15734237
- [Result] Shultz SJ, Sander TC, Kirk SE, Perrin DH. Sex differences in knee joint laxity change across the female menstrual cycle. J Sports Med Phys Fitness. 2005 Dec;45(4):594-603. PMID 16446695
- [Result] Dugan SA. Sports-related knee injuries in female athletes: what gives? Am J Phys Med Rehabil. 2005 Feb;84(2):122-30. doi: 10.1097/01.phm.0000154183.40640.93. PMID 15668560
- [Result] Demange MK, de Almeida AM, Rodeo SA. Updates in biological therapies for knee injuries: tendons. Curr Rev Musculoskelet Med. 2014 Sep;7(3):239-46. doi: 10.1007/s12178-014-9230-2. PMID 24957507
- [Result] Treatment of medial collateral ligament injuries of the knee with focused extracorporeal shockwave therapy: A case report.
- [Result] Moya D, Ramon S, Schaden W, Wang CJ, Guiloff L, Cheng JH. The Role of Extracorporeal Shockwave Treatment in Musculoskeletal Disorders. J Bone Joint Surg Am. 2018 Feb 7;100(3):251-263. doi: 10.2106/JBJS.17.00661. No abstract available. PMID 29406349
- [Result] Role of physiotherapy and physical agent modalities for musculoskeletal disorders: Present and future. Applied Sciences, 13(11), 6461
- [Result] Gesslbauer C, Mickel M, Schuhfried O, Huber D, Keilani M, Crevenna R. Effectiveness of focused extracorporeal shock wave therapy in the treatment of carpal tunnel syndrome : A randomized, placebo-controlled pilot study. Wien Klin Wochenschr. 2021 Jun;133(11-12):568-577. doi: 10.1007/s00508-020-01785-9. Epub 2020 Dec 22. PMID 33351153
- [Result] Ke MJ, Chen LC, Chou YC, Li TY, Chu HY, Tsai CK, Wu YT. The dose-dependent efficiency of radial shock wave therapy for patients with carpal tunnel syndrome: a prospective, randomized, single-blind, placebo-controlled trial. Sci Rep. 2016 Dec 2;6:38344. doi: 10.1038/srep38344. PMID 27910920
- [Result] Wang CJ. An overview of shock wave therapy in musculoskeletal disorders. Chang Gung Med J. 2003 Apr;26(4):220-32. PMID 12846521
- [Result] Wuerfel T, Schmitz C, Jokinen LLJ. The Effects of the Exposure of Musculoskeletal Tissue to Extracorporeal Shock Waves. Biomedicines. 2022 May 6;10(5):1084. doi: 10.3390/biomedicines10051084. PMID 35625821